CLINICAL TRIAL: NCT04613739
Title: Comparing Patient-Centered Outcomes for Adults and Children With Asthma in High-Deductible Health Plans With and Without Preventive Drug Lists: COVID Enhancement
Brief Title: Asthma in Families Facing Out-of-pocket Requirements Due to COVID-19
Acronym: AFFORD COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Asthma and Allergy Foundation of America (Other); University of North Carolina, Chapel Hill (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IHS-1602-34331
Record Dates: First submitted 2020-10-29; First posted 2020-11-03 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: health insurance; COVID-19; out-of-pocket health care costs; adherence; financial burden
MeSH Terms: conditions — Asthma; COVID-19; Financial Stress

STUDY DESIGN:
Masking Description: Outcomes will be assess through an online survey of participants with additional recoding done by an analyst blinded to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insurance navigation (Experimental): The intervention group will be offered access to AAFA's insurance chat bot and navigation services. Navigation will be provided through AAFA's existing online patient community platform that provides assistance with clinical, educational and financial questions and includes secure, personal messaging capabilities that will be supplemented with telephonic outreach.
  Interventions: Behavioral: insurance navigation
- Wait-list controls (No Intervention): Control subjects will be offered the chat bot after completion of data collection for the intervention group (after completion of the four-month follow-up surveys)

INTERVENTIONS:
Behavioral: insurance navigation — Intervention subjects will be offered access to AAFA's chat bot and navigation services. The chat bot is an artificial intelligence-enabled interactive online tool that can answer clinical and insurance-related questions and provide information on coverage options and how to find lower-cost alternatives for asthma care. Intervention participants will be given a link to access the chat bot. They will also be provided with information about AAFA's insurance navigation program, how it can help with finding coverage and managing asthma costs, and how to access it within AAFA's asthma community platform. Subjects can access AAFA's community platform and join the private group where they can ask questions and share resources, with moderation by AAFA staff. They will be able to send private messages to an AAFA navigator who can provide support about insurance issues, access to asthma care, and assistance with asthma costs. The navigator will offer telephonic follow-up as needed.
  Arms: Insurance navigation

SUMMARY:
In addition to its impact on health, the COVID-19 pandemic led to increased unemployment and loss of employer-sponsored insurance coverage. Obtaining coverage can be challenging and eligibility for public programs and subsidies can be limited, and those who do not qualify can face steep premiums, high-deductibles, and high out-of-pocket costs. Disruptions to employment and insurance coverage during the pandemic threaten to negatively affect asthma care and outcomes.

Our parent project, Asthma in Families Facing Out-of-pocket Requirements with Deductibles (AFFORD), found that patients with asthma may be particularly vulnerable to insurance-related cost barriers and challenges navigating health insurance. Together with the Asthma and Allergy Foundation of America (AAFA), the investigators developed an asthma chat bot to help patients with asthma navigate insurance benefits and optimize health care decisions. The chat bot is an artificial intelligence-enabled interactive online tool that can answer clinical and insurance-related questions and provide information on coverage and how to find lower-cost alternatives for asthma care.

In this supplement to the AFFORD project, the investigators propose a new study to understand and address the insurance and health care cost challenges faced by patients with asthma who lose employer-sponsored coverage due to COVID-19. Our Aims are: 1) to conduct a pilot randomized controlled trial to evaluate the effectiveness and feasibility and acceptability of an insurance navigation intervention, including the chat bot, to help patients with asthma regain coverage after the loss of job-related insurance during the COVID-19 pandemic; and 2) to qualitatively explore the experiences of Aim 1 participants to understand barriers and facilitators to accessing coverage and asthma care more broadly during the COVID-19 pandemic

The study hypothesis is that participants receiving the intervention will be more likely to have coverage after four months and less likely to report non-adherence to asthma medications, delayed/forgone asthma care, and financial burden than those receiving usual care. Findings will provide evidence about the effectiveness of strategies to obtain coverage and maintain access to affordable asthma care and can inform ongoing and future decision making in response to the COVID-19 pandemic and other public health and economic threats.

DETAILED DESCRIPTION:
In addition to its impact on health, the COVID-19 pandemic has led to increased unemployment and loss of employer-sponsored insurance coverage. Obtaining coverage can be challenging and eligibility for public programs and subsidies can be limited, and those who do not qualify can face steep premiums, high-deductibles, and high out-of-pocket costs. Disruptions to employment and insurance coverage during the pandemic threaten to negatively affect asthma care and outcomes.

Our parent project, Asthma in Families Facing Out-of-pocket Requirements with Deductibles (AFFORD), found that patients with asthma may be particularly vulnerable to insurance-related cost barriers and challenges navigating health insurance. Together with the Asthma and Allergy Foundation of America (AAFA), investigators developed an asthma chat bot to help patients with asthma navigate insurance benefits and optimize health care decisions. The chat bot is an artificial intelligence-enabled interactive online tool that can answer insurance-related questions and provide information on coverage and how to find lower-cost alternatives for asthma care.

In this supplement, the investigators propose to capitalize on the work of AFFORD to understand and address the insurance and health care cost challenges faced by patients with asthma who lose employer-sponsored coverage due to COVID-19. Specifically, our Aims are: 1) to conduct a pilot randomized controlled trial to evaluate the effectiveness and implementation outcomes (e.g. feasibility, acceptability) of an existing insurance navigation intervention, including the chat bot, to help patients with asthma regain coverage after the loss of job-related insurance during the COVID-19 pandemic; 2) to qualitatively explore the experiences of Aim 1 participants to understand barriers and facilitators to accessing coverage and asthma care more broadly during the COVID-19 pandemic

Findings will provide evidence about the effectiveness of patient-centered technological strategies to obtain coverage and maintain access to affordable asthma care and can inform ongoing and future decision making in response to the COVID-19 pandemic and other public health and economic threats.

Study Setting

Study participants will be recruited through the AAFA and Harvard Pilgrim Health Care. As in AFFORD, the proposed study will take advantage of AAFA's wide national reach and role as a trusted information source to recruit a national sample of patients with asthma or parents of children with asthma. We will also recruit through Harvard Pilgrim Health Care, a non-profit health plan that offers insurance plans in Massachusetts, Maine, New Hampshire, and Connecticut

Aim 1

In this aim, the investigators will conduct a pilot randomized controlled trial of patients with asthma or parents of children with asthma who lost employer-sponsored coverage during the COVID-19 pandemic. Potential study subjects will be recruited through AAFA and Harvard Pilgrim. Eligible participants will be randomized into one of two study groups: 1) an intervention group that receives access to an asthma chat bot and personalized insurance navigation (n=145), or 2) a wait-list control group (n=285). At study entry, participants will receive an online baseline survey to assess outcomes related to insurance coverage, asthma severity and control, medication use and adherence, asthma care access and affordability, and COVID-19 related illness. The intervention group will be offered the chat bot and AAFA navigation services. One month later, the investigators will field a follow-up survey to measure short-term changes in outcomes; for the intervention group, this survey will also measure implementation outcomes including uptake, feasibility, acceptability, and usability. Four months later, the investigators will field a second follow-up survey to measure longer-term changes in outcomes. Control subjects will be offered the chat bot after completion of the follow-up surveys.

Eligible subjects will include adults aged 18-64 years who have asthma or have a child with asthma aged 4-17 years, and lost employer-sponsored health insurance after February 2020. Potential subjects will be recruited through AAFA, who will send out a description of the study to potential subjects through its online community, email listserv, website, Facebook page, and newsletter. Potential subjects will also be recruited through Harvard Pilgrim. Members who disenrolled from employer-sponsored plans after February 2020 will be identified, and those aged 4-64 with an International Classification of Diseases (ICD)-10 diagnosis code for asthma in claims data after January 1, 2019 will be contacted by email and invited to participate. The investigators will collect information on race/ethnicity and select a sample representative of the racial/ethnic distribution of patients with asthma, with no more than 60% non-Hispanic White participants selected for the sample.

The investigators will conduct a pilot randomized controlled trial where they will randomize participants who lost coverage to: 1) be offered a combination of automated chat bot and personalized outreach provided by AAFA-affiliated navigators (n=145), or 2) be a wait-list control (n=285). The investigators will use a wait-list, usual care control group as the comparator given that there is no other standard treatment or practice for people with asthma who lose insurance coverage to which to compare our navigation intervention. After randomization, participants will be given a RedCap link for a baseline survey.

After completion of the baseline survey, intervention subjects will be sent an email with information about AAFA's asthma chat bot and a link to access it and information about AAFA's insurance navigation program, how it can help with finding coverage and managing asthma costs, and how to access it via group and private messaging within AAFA's asthma community platform with the availability of telephonic follow-up from AAFA navigators. Subjects can join the private group where they can ask questions and share resources. They will be able to send messages to the AAFA navigator to communicate about insurance issues, access to asthma care, and assistance with asthma costs. The navigator will offer telephonic follow-up as needed.

One month after receiving the intervention, subjects will be emailed a RedCap link to a follow-up survey to measure changes in insurance coverage and other outcomes. The follow-up survey will be structured similarly to the baseline survey, with closed-ended questions about insurance coverage, asthma care and control, health care access and affordability. For intervention subjects, the follow-up survey will also ask closed and open-ended questions about implementation outcomes such as uptake, acceptability, feasibility, usability, and fidelity.

Four months later, intervention and control subjects will be emailed a RedCap link to a similar follow-up survey to measure changes in insurance coverage, asthma care and control, health care access, and affordability. Survey subjects will be asked for permission to be contacted again for participation in a telephone interview for Aim 2.

The primary outcome will be whether the participant with asthma (or their child with asthma) has insurance coverage. Secondary outcomes will include whether the person with asthma used less asthma medication than prescribed because of cost, and whether they experienced health care-related financial burden. Other outcomes will assess asthma care use, asthma control using the Asthma Control Test (ACT), health status, mental health/worry, and material hardships such as food or housing insecurity.

The study hypothesis is that participants receiving the intervention will be more likely to have coverage at four-month follow up (primary outcome) and will be less likely to report non-adherence to asthma medications, delayed/forgone asthma care, and financial burden than those receiving usual care (secondary outcomes).

The investigators will compare unadjusted outcomes between the intervention and control groups using chi square and t tests; because of the randomized study design this difference measures the causal impact of the intervention. They will conduct post hoc exploratory analysis to assess differences in intervention effectiveness by race/ethnicity to assess whether the intervention reduces racial/ethnic coverage disparities. Given the small pilot nature of this study, these analyses will be hypothesis-generating rather than hypothesis-testing. In this pilot study, efficacy testing will be limited but the investigators expect to have 100 intervention and 200 control subjects with follow-up data to be able to detect absolute differences of 10% or more between study groups in changes in uninsurance rates with 80% power with a two-tailed alpha of 0.05. The investigators assume 30% loss to follow-up from baseline to four-month follow-up. Given the small pilot nature of this study, dropout will be carefully tracked in order to inform feasibility assessment and planning for a larger trial. The investigators will closely monitor timing of dropout, impact of strategies such as telephone outreach, and characteristics of those dropping out compared to those retained, and will use multiple imputation methods to conduct a sensitivity analysis to test the sensitivity of findings analyzed with and without imputed data. Findings will be reported using CONSORT reporting guidelines.

Aim 2

In this aim, the investigators will conduct in-depth qualitative interviews to better understand barriers and facilitators to accessing coverage and asthma care more broadly during the COVID-19 pandemic. Study subjects will be selected from among those who completed the follow-up survey and gave permission to be re-contacted for a telephone interview. The investigators will approach 100 eligible survey participants by email to invite them to participate in an interview. They expect to complete 30 phone interviews, half from the intervention group and half from the control group. Interviews will use open-ended questions to explore patients' experiences related to obtaining coverage after job loss and associated asthma care access and affordability challenges and facilitators. Interviews will be conducted by the study investigators and will be audio recorded and the recordings will be transcribed.

Eligible participants will be intervention and control participants who complete the four-month follow-up survey, give permission to be re-contacted for an interview, and provide an email and/or phone number to use to contact them. The investigators will seek to maximize variation in our sample by using survey data to identify potential subjects with a range of races/ethnicities, incomes, geographic residences, ages (child vs adult), and asthma severity.

The investigators will collect data from 30 study participants through in-depth qualitative interviews. They will approach 100 eligible survey participants by email to invite them to participate in an interview. They will then follow up by phone to schedule an interview. After scheduling a telephone interview and describing the study, they will obtain verbal informed consent. Interviews will last for approximately 45 minutes and will be audio recorded with permission and transcribed verbatim. They estimate completing 30 phone interviews, half with participants from the intervention group and half from the control group.

The investigators will transcribe recordings of the interviews and analyze these data via thematic content analysis. Using a codebook, 2 trained coders will independently code transcripts using NVivo, resolving disagreements via discussion. They will describe data thematically to probe quantitative findings and describe strengths, weaknesses, and perceived intervention impact.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* Adults aged 18-64 years who have asthma or have a child with asthma aged 4-17 years
* Lost employer-sponsored health insurance after COVID-19 was declared a pandemic in March 2020

Exclusion Criteria:

* Previous use of AAFA's insurance chat bot

Aim 2 (qualitative study):

As above, plus:

Inclusion Criteria:

- Completed four-month follow-up survey for Aim 1

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Galbraith, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insurance Navigation | Wait-list Controls
Started | 19 | 37
Completed (Completed four-month survey) | 12 | 25
Not Completed | 7 | 12
Not completed — Lost to Follow-up | 6 | 9
Not completed — potentially duplicative/fraudulent | 1 | 3

BASELINE CHARACTERISTICS:
Population: This is the number of participants randomized after completing the screening survey. Baseline characteristics come from the screening survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insurance Navigation | Wait-list Controls | Total
Number analyzed (Participants) | 19 | 37 | 56
Age, Customized [Count of Participants; unit: Participants]
  Age of reference patient (years): <=17 | 0 | 2 | 2
  Age of reference patient (years): 18-39 | 10 | 22 | 32
  Age of reference patient (years): 40-64 | 9 | 13 | 22
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender of reference patient: Male | 3 | 6 | 9
  Gender of reference patient: Female | 16 | 30 | 46
  Gender of reference patient: Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of reference patient
  Participants
    Hispanic or Latino | 3 | 4 | 7
    Not Hispanic or Latino | 15 | 31 | 46
    Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of reference patient
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 0 | 4 | 4
    White | 17 | 27 | 44
    More than one race | 0 | 4 | 4
    Unknown or Not Reported | 2 | 1 | 3
Recruitment source [Count of Participants; unit: Participants]
  Asthma and Allergy Foundation of America (AAFA) | 7 | 22 | 29
  Harvard Pilgrim | 12 | 15 | 27
Insurance status at baseline [Count of Participants; unit: Participants]
  Insured | 12 | 20 | 32
  Uninsured | 3 | 7 | 10
  Missing | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Insurance Coverage
Description: Coverage status (has any insurance coverage or not)
Time Frame: At follow-up (four months)
Measure: Count of Participants; unit: Participants
Arm/Group | Insurance Navigation | Wait-list Controls
Number analyzed (Participants) | 12 | 25
Participants
  Insured | 11 | 17
  Uninsured | 1 | 8

2. Secondary Outcome: Medication Adherence
Description: Report of using less asthma medication than prescribed because of cost
Time Frame: At follow-up (four months)
Measure: Count of Participants; unit: Participants
Arm/Group | Insurance Navigation | Wait-list Controls
Number analyzed (Participants) | 12 | 25
Participants
  Used less medication | 3 | 8
  Did not use less medication | 9 | 17

3. Secondary Outcome: Financial Burden
Description: Report of: 1) problems paying medical bills for asthma care, or 2) having to borrow money because of the amount required to pay for asthma care
Time Frame: At follow-up (four months)
Measure: Count of Participants; unit: Participants
Arm/Group | Insurance Navigation | Wait-list Controls
Number analyzed (Participants) | 12 | 25
Participants
  financial burden | 5 | 15
  no financial burden | 7 | 10

4. Secondary Outcome: Delayed/Forgone Care Due to Cost
Description: Change in report of: 1) using less asthma medication than prescribed because of cost,or 2) delaying or avoiding going to the doctor for asthma because of cost
Time Frame: From baseline to follow-up (four months)
Measure: Count of Participants; unit: Participants
Arm/Group | Insurance Navigation | Wait-list Controls
Number analyzed (Participants) | 12 | 25
Participants
  Delayed/forgone asthma care due to cost | 4 | 13
  No delayed/forgone asthma care due to cost | 8 | 12

ADVERSE EVENTS:
Time Frame: 8 months, 24 days
Arm/Group | Insurance Navigation | Wait-list Controls
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/37
Other Adverse Events (participants affected / at risk) | 0/19 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04613739/Prot_SAP_000.pdf